CLINICAL TRIAL: NCT03550157
Title: A Pilot Study of Cutaneous Ultrasound Evaluation of Structural Changes in Subcutaneous Tissue in Patients With Cellulitis After Multidisciplinary Treatment to Combat Cellulitis (PnKCelulitis® Program)
Brief Title: Structural Changes of Subcutaneous Tissue by Ultrasonographies in Patients After Treatment With PnKCelulitis® Program
Acronym: PnKCelulitis
Status: Completed | Type: Observational
Sponsor: Protein Supplies SL (Other)
Responsible Party: Sponsor
Other Study IDs: PNK-CEL-2016-06
Record Dates: First submitted 2018-05-08; First posted 2018-06-08 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2017-10

CONDITIONS: Cellulite
Keywords: Cellulite; Cutaneous ultrasound; PnKCelulitis® program
MeSH Terms: conditions — Cellulite

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 110 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Exploratory, prospective, uncontrolled and single-blinded pilot study, with clinical and ultrasound assessments of cutaneous cellulite before and after treatment with a specific multidisciplinary programme following dietary guidelines, physical exercise and the application of a cosmetic cream.

DETAILED DESCRIPTION:
Females older than 18, with normal weight ranges in addition to the presence of cutaneous non-infectious cellulite (edematous-fibrosclerotic panniculopathy), were recruited for the study and to undergo treatment with the multidisciplinary programme.

All patients were treated with the specific multidisciplinary programme for cellulite (PnKCelulitis®). This programme consists of three phases or processes: the restructuring, drainage and toning processes, each of which combines diet, physical exercise and the application of an anti-cellulite cream that combines active lipolytic and vasodilator agents (Cellulite Gel K-Line®).

Patient's clinical assessment follow-up was performed by the prescribing doctor for the multidisciplinary treatment and was done in four visits: baseline (before starting treatment) and at the end of each of the phases (restructuring, drainage and toning). Anthropometric data were recorded at each visit and a bioelectric impedance test to assess body composition (amount of fat mass and muscle mass). The clinical evaluation of the degree of cellulite was made according to the Nürnberger-Muller classification scale.

Cutaneous ultrasound was performed by an expert dermatologist in the dermatology outpatient clinic of the hospital and subsequently assessed blinded. Two skin scans were done for each patient, one before starting the treatment and another at the end. The objective data collected on each ultrasound were total skin thickness, thickness of the dermis and hipodermis, the area of the indentations of the subcutaneous cellular tissue in the dermis and changes in the echogenicity of the dermis blinded and independently assessed by two researchers, comparing ultrasounds before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Females older than 18 years
* Normal weight ranges
* Presence of cutaneous non-infectious cellulite (edematous-fibrosclerotic panniculopathy)
* Women who are going to begin treatment with the multidisciplinary programme

Exclusion Criteria:

* Pregnant or lactating females
* Contraindications of a ketogenic diet

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cellulite or edematofibrosclerotic panniculopathy is a disorder that affects 85-98% of females after puberty and is considered a secondary sexual trait in females
Study Population: Females older than 18, with normal weight ranges in addition to the presence of cutaneous non-infectious cellulite (edematous-fibrosclerotic panniculopathy), were recruited for the study and to undergo treatment with the multidisciplinary programme.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-09-27 (Actual); Primary Completion 2017-01-30 (Actual); Study Completion 2017-04-26 (Actual)

PRIMARY OUTCOMES:
Thickness of the hypodermis reduction | from the beginning to the end of treatment, an average of 8±1 weeks in patients with grade 1, an average of 10±1 weeks in patients with grade 2 and an average of 14±1 weeks for patients with grade 3
  Change in thickness of the hypodermis reduction measured by cutaneous ultrasound from baseline to end of treatment
Area of indentations reduction | from the beginning to the end of treatment, an average of 8±1 weeks in patients with grade 1, an average of 10±1 weeks in patients with grade 2 and an average of 14±1 weeks for patients with grade 3
  Change in area of the indentations of the subcutaneous cellular tissue in the dermis from baseline to end of treatment measured by cutaneous ultrasound

SECONDARY OUTCOMES:
Total skin thickness reduction | from the beginning to the end of treatment, an average of 8±1 weeks in patients with grade 1, an average of 10±1 weeks in patients with grade 2 and an average of 14±1 weeks for patients with grade 3
  Change in total skin thickness measured by cutaneous ultrasound from baseline to end of treatment
Thickness of dermis reduction | from the beginning to the end of treatment, an average of 8±1 weeks in patients with grade 1, an average of 10±1 weeks in patients with grade 2 and an average of 14±1 weeks for patients with grade 3
  Change in total thickness of dermis measured by cutaneous ultrasound from baseline to end of treatment
Cellulite grade reduction | from the beginning to the end of treatment, an average of 8±1 weeks in patients with grade 1, an average of 10±1 weeks in patients with grade 2 and an average of 14±1 weeks for patients with grade 3
  Change in the degree of cellulitis according to the Nürnberger-Muller classification scale from the beginning to the end of the treatment. It is a simple grading-score of cellulite by inspection (grade 0= Smooth surface of skin while lying down and standing and wrinkles upon pinch-test; grade 1=Smooth surface of skin while lying down and standing, mattress-phenomenon upon pinch-test; grade 2=Mattress-phenomenon spontaneously while standing and grade 3=Mattress-phenomenon spontaneously while standing and lying down). A higher score indicates a higher severity of cellulite.
Body weight reduction | from the beginning to the end of treatment, an average of 8±1 weeks in patients with grade 1, an average of 10±1 weeks in patients with grade 2 and an average of 14±1 weeks for patients with grade 3
  Change in body weight from baseline to end of treatment
Body Mass Index reduction | from the beginning to the end of treatment, an average of 8±1 weeks in patients with grade 1, an average of 10±1 weeks in patients with grade 2 and an average of 14±1 weeks for patients with grade 3
  Change in Body Mass Index from baseline to end of treatment
Skeletal muscle mass increase | from the beginning to the end of treatment, an average of 8±1 weeks in patients with grade 1, an average of 10±1 weeks in patients with grade 2 and an average of 14±1 weeks for patients with grade 3
  Change in skeletal muscle mass from baseline to end of treatment
Body fat mass reduction | from the beginning to the end of treatment, an average of 8±1 weeks in patients with grade 1, an average of 10±1 weeks in patients with grade 2 and an average of 14±1 weeks for patients with grade 3
  Change in body fat mass from baseline to end of treatment
Abdominal perimeter reduction | from the beginning to the end of treatment, an average of 8±1 weeks in patients with grade 1, an average of 10±1 weeks in patients with grade 2 and an average of 14±1 weeks for patients with grade 3
  Change in abdominal perimeter (navel level) from baseline to end of treatment
Low abdominal perimeter reduction | from the beginning to the end of treatment, an average of 8±1 weeks in patients with grade 1, an average of 10±1 weeks in patients with grade 2 and an average of 14±1 weeks for patients with grade 3
  Change in low abdominal perimeter (5 cm below navel) from baseline to end of treatment
Thigh perimeter reduction | from the beginning to the end of treatment, an average of 8±1 weeks in patients with grade 1, an average of 10±1 weeks in patients with grade 2 and an average of 14±1 weeks for patients with grade 3
  Change in thigh perimeter from baseline to end of treatment
Number of Participants With Adverse Events | from the beginning to the end of treatment, an average of 8±1 weeks in patients with grade 1, an average of 10±1 weeks in patients with grade 2 and an average of 14±1 weeks for patients with grade 3
  Number of Participants With Adverse Events as a Measure of Safety and Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Esther Roe, Ph, Principal Investigator — Hosptial de al Santa Creu i Sant pau

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-05): https://cdn.clinicaltrials.gov/large-docs/57/NCT03550157/Prot_SAP_000.pdf